CLINICAL TRIAL: NCT03162237
Title: Investigation of Safety and Efficacy Study of Islets Xenotransplantation for Patients With Type 1 Diabetes
Brief Title: Safety and Efficacy Study of Islets Xenotransplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wei Wang,MD (Other)
Collaborators: Hunan Xeno-life Science Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Wei Wang,MD, Director of Cell Transplantation and Gene Therapy Institute, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CellTransplant&GeneTherapy2013
Record Dates: First submitted 2014-01-29; First posted 2017-05-22 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Type 1 Diabetes
Keywords: Type1 diabetes; porcine islets; treg cells; immunosuppress; xenotransplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Porcine islets and autologous treg (Experimental): Porcine islets:10000 islet equivalent（IEQ）/Kg; Treg:2x10^6/Kg
  Interventions: Other: Porcine islets; Other: Autologous Treg
- AutologousTreg (Active Comparator): Autologous Treg:2x10^6/Kg
  Interventions: Other: Autologous Treg

INTERVENTIONS:
Other: Porcine islets — Porcine islets: 10000IEQ/Kg;
  Tacrolimus: 0.087mg/kg, Bid;
  mycophemo-latemofetil (MMF): 1g x 2/d;
  NULOJIX(belatacept): Day 1 (prior to transplantation), Day 5, Week 2, Week 4, Week 8, Week 12 10mg/kg
  Arms: Porcine islets and autologous treg
Other: Autologous Treg — Autologous Treg: 2x10^6/Kg

SUMMARY:
The neonatal pig islets will be used as donor culturing with our modified culture medium. At the same time the autologous T regulatory cells will be used to induce specific immune tolerance for porcine islets grafts combined the costimulation of T cell activation channel blockers. The treatment for type 1 diabetes will be evaluated the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 40 years of age;
* Type 1 diabetes mellitus for at least 5 years;
* Body weight 40 to 60kg;
* Ability to provide written informed consent;
* Manifest signs and symptoms that are severe enough to be incapacitating;
* Patients with poor diabetes control (HbA1c > 9% );
* Patients have diabetes ketoacidosis or hypoglycemia more than once

Exclusion Criteria:

* Age < 18 years or > 60 years;
* Diabetes history < 5 years;
* Body weight > 80 kg;
* Exogenous insulin requirement > 1 unit/kg/day;
* Blood test: hemoglobin male < 90g/l, female < 90 g/l) or Wbc <3×109/L, lymphocyte <1.5×10^9/L; or platelet < 80×10^9/L; activated- partial-thromboplastin-time （APTT） > normal value (31-43s)10s;
* Liver dysfunction;
* Kidney dysfunction;
* Cardiopulmonary dysfunction;
* Combined mental illness, cancer, infection, severe trauma, pancreatitis, surgery or other stress situations for patients; gastric ulcer patients, any bleeding disorders, tuberculosis infection and active infection including hepatitis B, hepatitis C, HIV, or John Cunningham virus;
* Serological detection Epstein-Barr virus (EBV) or Cytomegalovirus (CMV)negative;
* Patient have taken immunosuppressant in recent one year With high incidence of malignancy in three generation;
* Women not using effective contraception of childbearing age, or planning pregnancy in nearly two years or being pregnant or lactating;
* Patients can not comply with the research program to complete the diagnosis and treatment;
* Patients not be passed by Ethics committee

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose | 1 year
  Before and after transplantation the patient will be tested the blood glucose. If the blood glucose within 24 hours is stable and no occurrence of diabetic ketoacidosis and hypoglycemia.Thirty percent reduction of exogenous insulin requirement will be considered as effective.

SECONDARY OUTCOMES:
Porcine C-peptide | 1 years
  The patient will be detected the porcine C-peptide levels after transplantion every three months.
Hemoglobin A1c | 1 years
  After transplantation the patient will be checked hemoglobin A1c every month.The level of HbA1c less than 6.5% was considered as effective.
AST | 1 years
  AST will be tested every three months.
ALT | 1 years
  ALT will be tested every three months.
Scr | 1 years
  Scr will be tested every three months.
BUN | 1 years
  BUN will be tested every three months.
Ultrasonic examination for liver | 1 years
  Ultrasonic examination will be used for the recipient's liver before transplantation and every three month post transplantation.
MRI for liver | 1 years
  MRI will be used for liver before transplantaion and every three month post transplantation.
Virus detection | 2 years
  The recipient's serum and peripheral blood monouclear cells (PBMC) will be collected for virus detection every six months.
Immune cells detection | 1 years
  The recipient's peripheral blood monouclear cells (PBMC) and the serum will be collected for immune cell's analysis.
Cytokine detection | 1 years
  The recipient's peripheral blood monouclear cells (PBMC) and the serum will be collected cytokine beads array (CBA) test.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PHD,MD, Study Chair — Cell transplantation and gene therapy, the 3rd Xiangya hospital of Central South University
Locations (1):
- Cell Transplantation and Gene Therapy Institute, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No